CLINICAL TRIAL: NCT05062174
Title: Targeting Progesterone Signaling for Breast Cancer Prevention in BRCA1 Carriers: a Pilot Study
Brief Title: Breast Cancer BRCA1 Carriers: a Pilot Study
Status: Withdrawn | Type: Observational
Why Stopped: PI decision to cancel research
Sponsor: Indiana University (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor Clinical Medicine, Indiana University
Other Study IDs: CTO-IUSCCC-0758
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: BRCA1 Mutation; High-grade Serous Ovarian Cancer; TNBC - Triple-Negative Breast Cancer
Keywords: progesterone signaling; mifepristone; glucocorticoid receptor; androgen receptor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — Mifepristone; Prophylactic Mastectomy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — random core biopsy of breast tissue from one breast at time of biopsy and pre-planned mastectomy, as well as blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mifepristone + surgery: Mifepristone is taken orally as a one-time only dose between 48 and 56 hours before your planned prophylactic mastectomy surgery
  Interventions: Drug: Mifepristone 200 MG; Procedure: Prophylactic mastectomy

INTERVENTIONS:
Drug: Mifepristone 200 MG — Orally, one time dosage of 200 mg
Procedure: Prophylactic mastectomy — Planned prophylactic mastectomy (having one or both breasts removed).

SUMMARY:
The purpose of this study is to examine how a single dose of MIFEPREX® (mifepristone) affects the breast tissue in patients with BRCA1 (a gene that normally acts to restrain the growth of cells in the breast, but if it mutates may lead to breast cancer) mutations undergoing a planned prophylactic mastectomy (having one or both breasts removed).

DETAILED DESCRIPTION:
This is a single arm, prospective, observational trial enrolling up to 10 patients within Indiana University Simon Comprehensive Cancer Center. Eligible women will be consented to undergo breast biopsy 2-6 days prior to prophylactic mastectomy and take one dose of mifepristone 2 days prior to prophylactic mastectomy. If the initial biopsy is obtained on Day -2, the mifepristone should be taken AFTER the biopsy. Tissue from the ipsilateral breast will be taken at the time of mastectomy.

Primary Objective To determine the impact of a single 200 mg dose of mifepristone on gene expression and metabolomic alterations in breast tissue of women with BRCA1 mutations who are planning prophylactic mastectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 old at the time of informed consent
2. Known pathogenic germline BRCA1 mutation. The mutation must have been discovered by a CLIA- approved next generation sequencing panel (such as Myriad, Invitae, Ambry, etc) and confirmed by the PI.
3. Planning to undergo prophylactic risk reducing mastectomy
4. Premenopausal, defined as:

   1. At least one ovary remains in situ, AND
   2. Estradiol > 20 or last menstrual period within the prior 3 months
   3. Prior hysterectomy is allowed as long as at least one ovary remains in place
5. Must not be pregnant or nursing

   a. Must have a negative urine pregnancy test for registration and between -6 to day -2 prior to receiving mifepristone
6. Ability to provide written informed consent and HIPAA authorization
7. Agrees to pre-treatment core biopsy with donation to the IUSCCC Komen Normal Tissue Bank. Patient will sign a separate informed consent for donation to the IUSCCC Komen Normal Tissue Bank.

Exclusion Criteria:

1. Patients may not have used progesterone-only contraceptives (i.e. Depo- Provera) within the last 6 months. Combination estrogen/progesterone or estrogen only contraceptives are allowed.
2. Presence of an intrauterine device
3. Personal history of breast or ovarian cancer
4. Active heavy smoker, defined as 10 or more cigarettes per day on any occasion in the past 30 days
5. Uncontrolled chronic medical condition, including insulin dependent diabetes, NYHA class II, III or IV congestive heart failure, unstable angina, history of myocardial infarction, chronic pulmonary conditions including uncontrolled asthma (symptoms > 2 days/week) or dyspnea requiring oxygen, peripheral vascular disease, symptomatic anemia, uncontrolled psychiatric conditions, chronic kidney disease, or liver disease (cirrhosis, NAFLD, etc.)
6. Requiring ongoing therapy with strong CYP3A4 inhibitor, steroids, or immunosuppressants (i.e. tacrolimus, cyclosporine, etc.). Please see appendix for full list of excluded co-medications. If questions, please ask the PI.
7. History of life- threatening allergic reaction to local anesthesia (lidocaine, xylocaine).
8. Contraindications including but not limited to allergic reactions to mifepristone or other prostaglandins, or inherited porphyrias
9. For the purposes of invasive breast biopsies, women must not be receiving therapeutic anticoagulation or antiplatelet agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 BRCA-1 mutation carriers who plan to undergo prophylactic mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of mifepristone | From baseline (day -2 to day -6) to Breast surgery (day 0)
  To determine the impact of a single 200 mg dose of mifepristone on gene expression and metabolomic alterations in breast tissue of women with BRCA1 mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana